CLINICAL TRIAL: NCT04066335
Title: An Observational Study to Evaluate the Safety of Nanoxel M (Docetaxel-PM) Inj.
Brief Title: Study to Evaluate the Safety of Nanoxel M Inj.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DPM401
Record Dates: First submitted 2019-08-14; First posted 2019-08-26 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Non-small Cell Lung Cancer; Prostate Cancer; Ovarian Cancer; Head and Neck Cancer; Gastric Cancer; Esophageal Cancer
Keywords: Observational Study, Safety, Nanoxel M, Docetaxel
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Ovarian Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study to evaluate the safety of Nanoxel M inj. administration in patients.

DETAILED DESCRIPTION:
This is a multi-center, prospective observational study to observe the incidence of adverse events under actual clinical settings to test the safety of Nanoxel-M inj. administration in patients with breast cancer, non-small cell lung cancer, prostate cancer, ovarian cancer, head & neck cancer, gastric cancer or esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years old
2. Patients who have signed written consent form prior to participating in the clinical trial
3. Patients who are assessed as adequate to administer Nanoxel M injection.

Exclusion Criteria:

1) Patients who have shown severe hypersensitivity to Docetaxel and concomitant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are assessed as adequate to administer Nanoxel M inj.
Sampling Method: Non-Probability Sample
Enrollment: 1498 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Safety of Nanoxel M inj. | through study completion, an average of 6cycles(each cycle is 3weeks)
  The incidence of Treatment-Emergent Adverse Event

CONTACTS AND LOCATIONS:
Locations (1):
- Samyang Biopharmaceuticals, Seoul, South Korea